CLINICAL TRIAL: NCT01371435
Title: Drug Use Investigation for PAXIL Tablet
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112301
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Paroxetine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients prescribed PAXIL: Patients with depression/depressed state or panic disorder prescribed PAXIL during study period
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
This post-marketing surveillance study is designed to detect adverse events (particularly clinically significant adverse drug reactions) occurring in clinical settings and to examine factors likely to affect the safety and efficacy of paroxetine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with depression/depressed state or panic disorder

Exclusion Criteria:

* Patients who had been taking PAXIL since before the start of the survey
* Patients with hypersensitivity to paroxetine
* Patients taking monoamine oxidase inhibitors (MAOIs) or within 2 weeks of stopping treatment with MAOIs
* Concomitant use in patients taking pimozide

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with depression/depressed state or panic disorder who were indicated for PAXIL
Sampling Method: Probability Sample
Enrollment: 3708 (Actual)
Dates: Start 2001-04; Primary Completion 2005-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in Japanese subjects treated with paroxetine tablet based on prescribing information under the conditions of general clinical practice | 8 weeks
Presence/absence of concomitant use of drugs metabolized by CYP2D6 | Within 2 weeks after discontinuation or completion of treatment
  PAXIL inhibits drug-metabolizing enzyme CYP2D6, and it takes about 1 week following discontinuation of PAXIL for this CYP2D6 function to recover from the inhibiting effect. Since it requires attention if drugs that are metabolized by CYP2D6 are administered during this recovery period, it was decided to investigate the presence/absence of use of drugs metabolized by CYP2D6 within 2 weeks after discontinuation of treatment in patients for whom treatment with PAXIL was discontinued, as well as the safety thereof.
Presence/absence of concomitant use of products containing Saint John's Wort (Hypericum perforatum; "SJW", hereinafter) | 8 weeks
  Although the action mechanism for this is not clear, SJW has been reported to have the action of inhibiting reuptake of serotonin, noradrenaline and dopamine, and to exhibit an antidepressant effect. Since PAXIL also acts to inhibit serotonin reuptake, concomitant use of products containing SJW is thought to have an effect upon the serotonin reuptake inhibiting action of PAXIL, so it was decided to check for concomitant use of products containing SJW and investigate the safety of such concomitant use.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline